CLINICAL TRIAL: NCT05570968
Title: Outcomes of Endovascular Revascularization in Patients With Chronic Limb Threatening Ischemia (CLTI) Associated With Heel Ulcers
Brief Title: Outcomes of Endovascular Revascularization in CLTI in Patients Associated With Heel Ulcers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yehia Mohamed Mostafa Abdelhadi, Resident, Assiut University
Other Study IDs: Endovascular revascularization
Record Dates: First submitted 2022-09-30; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Lower Limb Ischemia Critical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: C-arm device — Percutaneous Transluminal Angioplasty

SUMMARY:
The aim of the current study is to assess outcomes of endovascular revascularization of patients with CLTI associated with heel ulcers and identify possible predictors of healing of these ulcers.

DETAILED DESCRIPTION:
Peripheral Arterial Disease (PAD) is a progressive disorder characterized by stenosis and/or occlusion of large and medium-sized arteries and affects the lower extremities more commonly than the upper extremity vessels, and may lead to a recurrent fatigue, cramping sensation, or pain that is known as intermittent claudication, which is the most recognized symptomatic subset of lower extremity PAD. (1) Chronic limb threatening ischemia (CLTI) is an advanced form of PAD encompassing rest pain, lower limb ulceration or gangrene. It is associated with significant morbidity, mortality and healthcare resource utilization. (2) The Society for Vascular Surgery (SVS) Lower Extremity Guidelines Committee realized there was a need for a classification system for threatened limbs that encompassed the full spectrum of disease, as all existing classification systems fell short in this regard. So, they created the WIfI (Wound, Ischemia, and foot Infection) Classification System to categorize these three major risk factors leading to amputation. (3) It contains the key limb status elements needed to gauge the severity of limb threat, which enables physicians to predict amputation risk more accurately. (4) Either surgical or endovascular revascularization is the mainstay of therapy for CLTI. The continuous advance in the field of vascular interventional radiology has facilitated angioplasty through the development of low-profile balloon catheters, various small calibre stents, steerable and hydrophilic guide wires, road map facilities, vasodilators, and antiplatelet medication. (5) Heel ulcers in patients with diabetes mellitus (DM) and PAD are hard to heal. Diabetic heel ulcer is a well-known, hard to-heal ulcer and is considered a major risk factor for lower extremity amputation. Presence of foot ischemia, peripheral neuropathy with external trauma, and foot deformities will further increase the risk of amputation, and it is therefore highly likely that a patient with a diabetic heel ulcer with ischemia will have a great benefit from revascularization, especially if together with adequate infection control. (6)

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from CLTI associated with heel ulcers who will undergo endovascular revascularization at Assiut university vascular surgery department between August 2022 and November 2023.

Exclusion Criteria:

* Patients with arterial thrombosis , dissection, or embolism.
* Known intolerance to the study medications or contrast agents
* Patients with failing or failed bypass grafts

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with chronic limb threatening ischemia associated with heel ulcers Males or Females
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Treatment success | 1 year
  residual diameter stenosis of less than 30% at the end of the procedure as demonstrated on completion angiography
Procedural complications | 1 year
  according to the society of intervention radiology (SIR) criteria.

SECONDARY OUTCOMES:
Primary patency | 1 year
  freedom from clinically driven target lesion revascularization (CD-TLR) and restenosis (DUS peak systolic velocity ratio >2.5
CD-TLR | 1 year
  any re-intervention at the target lesion(s) due to symptoms or drop of ABI of ≥20% or >0.15 when compared to post-procedure baseline ABI
Amputation free survival (AFS) | 1 year
  s time until a major (above-ankle) amputation of the index limb or death from any cause.

REFERENCES:
- [Background] Butt T, Lilja E, Orneholm H, Apelqvist J, Gottsater A, Eneroth M, Acosta S. Amputation-Free Survival in Patients With Diabetes Mellitus and Peripheral Arterial Disease With Heel Ulcer: Open Versus Endovascular Surgery. Vasc Endovascular Surg. 2019 Feb;53(2):118-125. doi: 10.1177/1538574418813746. Epub 2018 Nov 22. PMID 30466379
- [Background] Linn YL, Chan SL, Soon SXY, Yap CJQ, Lim MNHH, Lee QWS, Chong TT, Tang TY. Heal or no heel: Outcomes of ischaemic heel ulcers following lower limb revascularization from a multi-ethnic Asian Cohort in Singapore. Int Wound J. 2020 Dec;17(6):2010-2018. doi: 10.1111/iwj.13493. Epub 2020 Aug 24. PMID 32840061